CLINICAL TRIAL: NCT06101316
Title: A Bridging Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of CB06-036 in Healthy Subjects in China
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhimeng Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CB06-036-102A
Record Dates: First submitted 2023-09-20; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CB06-036 Cohort 1 (Experimental): 1.5 mg Day1, orally taken in the morning, on an empty stomach.
  Interventions: Drug: CB06-036

INTERVENTIONS:
Drug: CB06-036 — CB06-036 Capsule

SUMMARY:
CB06-036 is an investigational drug developed by Shanghai Zhimeng Biopharma Inc. for the treatment of Chronic Hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide signed informed consent to participate in the study and understand the study content, procedures, and possible adverse reactions.
2. Able to finish the study in accordance with the study protocol.
3. Subjects (including partners) are willing to voluntarily take effective contraceptive measures within 6 months from screening until the last dose of the study drug (see Appendix 4 for specific contraceptive measures)
4. Male or Female, of age ≥18 and ≤50 years.
5. Body weight ≥50.0 kg for males and ≥45.0 kg for females, with BMI ≥ 18 and ≤ 28 kg/m2, BMI ＝ Body Weight (kg) / Height 2(m2).
6. No clinically significant abnormal finding on vital signs or physical examination at screening.
7. Estimated Glomerular Filtration Rate (eGFR) ≥ 60 mL/min calculated using the Modification of Diet in Renal Disease (Cockcroft-Gault MDRD) equations (see Appendix 6 for the details);
8. Liver function tests within the normal range for alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, and total bilirubin at screening.

Exclusion Criteria:

1. Having had major trauma or underwent major surgery within 3 months before screening.
2. With previous treatment, which may affect drug absorption (such as subtotal gastrectomy).
3. History of blood donation or massive blood loss (> 450 mL) within 3 months before screening.
4. Suspected of having a history of allergy to any ingredient of the study drug or allergic constitution (multiple drug and food allergy).
5. Smoked more than 5 cigarettes per day within 1 month before screening.
6. History of drug abuse and/or alcohol abuse (alcohol use exceeds 14 units per week; 1 unit = 285 mL of beer, or 100 mL of wine, or 25 mL of distilled alcohol).
7. Acute infections within 14 weeks before screening.
8. Clinically significant abnormalities on clinical laboratory tests or other clinical findings within 6 months prior to screening that indicates clinically significant disease of the following (including, but not limited to, gastrointestinal, renal, hepatic, neurological, hematological, endocrine, oncological, pulmonary, immunological, psychiatric, or cardiovascular disease);
9. Have known or historically documented uveitis, systemic lupus erythematosus, rheumatoid arthritis, psoriasis, Sjogren's syndrome, scleroderma, and other autoimmune diseases.
10. Have known or documented history of clinically significant fundus lesions (symptomatic fundus cotton-wool-spots) and retinopathy;
11. Have a known or documented history of clinically significant thyroid disease;
12. History of myocardial infarction, unstable angina, percutaneous coronary intervention (PCI), coronary artery bypass grafting (CABG), Grade III or IV heart failure, or stroke within 6 months before screening.
13. Plan to have surgery or be hospitalized during the study.
14. Have used immunosuppressants, immunomodulators (thymosin), and cytotoxic drugs within 6 months before screening;
15. Use of a class of drugs with a defined action that serves as moderately potent inhibitors or strong inducers, which can alter the activity of drug-metabolizing enzymes, etc., within 14 days before screening;
16. Have used any prescription drugs, over-the-counter drugs, vitamins, herbal or other diet or supplement deemed inappropriate by the Investigator within 7 days prior to screening;
17. Those who have been vaccinated within 14 days prior to screening or plan to be vaccinated during the study;
18. Those who have consumed a special diet (including dragon fruit, mango, grapefruit, etc.) or exercised vigorously within 3 days before screening, or have other factors that affect drug absorption, distribution, metabolism, excretion, etc.;
19. Having had chocolate, caffeine or xanthine-rich food or beverage, or any alcohol products 48 hours before study drug administration.
20. Have acute illness or using concomitant medication from screening to study drug administration;
21. Have had any investigational medicine or participated in the clinical study of medical devices within 3 months before screening.
22. With clinically significant ECG abnormalities judged by the investigator as not suitable for study participation.
23. Women of breast-feeding or with positive pregnancy test.
24. Positive screening for any of Hepatitis B serological test, hepatitis C[HCV] antibodies, Human immunodeficiency Virus[HIV], or Syphilis test.
25. Positive urine drug screen (morphine, marijuana) or alcohol breath test.
26. Have other factors that are not suitable for study participation in the investigator's opinion.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-29 (Estimated)

PRIMARY OUTCOMES:
Abnormalities of vital signs (blood pressure, pulse rate, temperature, and respiration rate) | At Screening，Baseline，Day1，Day 3
  Vital signs safe reference range:systolic blood pressure 84-139 mmHg, diastolic blood pressure 50-89 mmHg, pulse rate 50-100 times per min, temperature 35.9-37.6℃, respiration rate 12-20 times per min
Abnormalities of physical examination | At Screening，Baseline，Day 3
  Medical examinations performed by physicians include:Skin, mucous membranes, lymph nodes, head, neck, chest, abdomen, spine and limbs, nervous system
Abnormalities of 12-lead ECG | At Screening，Baseline，Day1，Day 3
  An ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTcF intervals should be used. Changes in T-wave, U-wave morphology and overall ECG interpretation will be documented.
Abnormalities of clinical laboratory | At Screening，Baseline，Day 3
  The clinical laboratory items includes：Blood routine, blood biochemistry, urine routine, blood clotting function, A function three, C Reactive protein
Abnormalities of Ophthalmic Examination | At Screening，Baseline，Day 3
  Ophthalmic examinations will be performed to assess ophthalmologic findings, including direct/indirect ophthalmologic examination, slit lamp and fundoscopic examination with retinal photographs (both eyes).Photographs of the retina must be taken.
Measure time of the maximum observed concentration 【Tmax】 | From 0.5 hour pre-dose to 24 hours post-dose
  To evaluate whether there are differences in the pharmacokinetic characteristics of CB06-036 in healthy subjects in China and the United States
Measure maximum observed concentration【Cmax】 | From 0.5 hour pre-dose to 24 hours post-dose
  To evaluate whether there are differences in the pharmacokinetic characteristics of CB06-036 in healthy subjects in China and the United States
Measure apparent terminal elimination half-life【t1/2】 | From 0.5 hour pre-dose to 24 hours post-dose
  To evaluate whether there are differences in the pharmacokinetic characteristics of CB06-036 in healthy subjects in China and the United States
Measure area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC0-∞) | From 0.5 hour pre-dose to 24 hours post-dose
  To evaluate whether there are differences in the pharmacokinetic characteristics of CB06-036 in healthy subjects in China and the United States
Measure area under the plasma concentration-time curve from the first dose to the last measurable sample collection time t (AUC 0-t) | From 0.5 hour pre-dose to 24 hours post-dose
  To evaluate whether there are differences in the pharmacokinetic characteristics of CB06-036 in healthy subjects in China and the United States
Measure Clearance (CL/F) | From 0.5 hour pre-dose to 24 hours post-dose
  To evaluate whether there are differences in the pharmacokinetic characteristics of CB06-036 in healthy subjects in China and the United States
Measure apparent volume of distribution (Vz/F) | From 0.5 hour pre-dose to 24 hours post-dose
  To evaluate whether there are differences in the pharmacokinetic characteristics of CB06-036 in healthy subjects in China and the United States

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zhang, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China